CLINICAL TRIAL: NCT03695042
Title: The Utilization of Blood Flow Restriction Training in Post Concussion Recovery
Brief Title: Blood Flow Restriction Concussion
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty enrolling target population within target timeframe
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Pro00100185
Record Dates: First submitted 2018-10-02; First posted 2018-10-03 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Concussion Post Syndrome
MeSH Terms: conditions — Post-Concussion Syndrome | interventions — Blood Flow Restriction Therapy; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BFR THEN without BFR (Experimental): Will perform exercises with BFR at the first visit and without BFR at the second visit
  Interventions: Other: Blood Flow Restriction Training with Exercise
- Without BFR THEN with BFR (Experimental): Will perform exercises without BFR at the first visit and with BFR at the second visit
  Interventions: Other: Blood Flow Restriction Training with Exercise

INTERVENTIONS:
Other: Blood Flow Restriction Training with Exercise — The addition of BFR training to an exercise program prescribed for a patient participating in physical therapy for concussion treatment. BFR training partially occludes blood flow to extremities during exercise. This allows one to exercise at lower loads and still gain benefits similar to exercise at higher loads

SUMMARY:
The purpose of this study is to examine the effect that blood flow restriction training will have on patients with concussion who demonstrate an intolerance to physical activity. Progressive exercise training has been shown to effectively reduce the effects of concussion and facilitate return to academic and athletic activities. In many cases, exercises intolerance is present in these patients which hinders progression. In musculoskeletal conditions, blood flow restriction training, when combined with low load exercise, has been shown to produce similar gains as high load exercises. If a patient being treated for concussion can tolerate low load exercise without concussive symptoms, then blood flow restriction may increase exercise gains by facilitating autonomic responses similar to high load training. This study will explore this hypothesis in patients between the ages of 14 and 30 who are referred for physical therapy intervention which is the standard of care at Duke Sports Sciences Concussion Clinic. Blood flow restriction training is also used in multiple patient populations at Duke Sports Physical Therapy without adverse events.

DETAILED DESCRIPTION:
This is a prospective randomized proof of concept trial comparing the efficacy of the novel application of blood flow restriction to improve exercise tolerance in patients with post-concussion syndrome. Blood flow restriction training is commonly used in combination with low intensity/load exercise to facilitate exercise tolerance in those that would not tolerate high intensity/load exercises. While this intervention has been clinically employed in patients with concussion, research is needed to establish it's efficacy in a meaningful and prospective way. Subjects in this study will be randomly assigned to one of two groups. One group will perform exercises with BFR and then without BFR. The other group will perform the exercises without BFR first and then perform them with BFR. Each subject will undergo a single physical therapy session in each condition. Subjects meeting study criteria will be randomly allocated to each group. Because concussion symptoms can change quickly over time, it will be important to vary the timing of when the blood flow restriction is performed to better understand if improvement is due to intervention or passage of time. Randomization will be performed via sealed envelope to ensure even distribution into both groups.

Patients presenting to physical therapy for treatment of concussion symptoms will undergo a physical therapy concussion evaluation that includes orthostatic measurements, cervical screen, and vestibular-oculomotor screen. Patients will report a Global Function Rating and complete a Post-concussion Symptom Score, Neck Disability Index, and Dizziness Handicap Inventory at initial visit. Heart rate variability will also be assessed at initial visit. The measurements and questionnaires collected at the initial evaluation are part of the standard of care at this clinic. Subjects will be recruited after the initial visit and will have already completed these measurements/questionnaires. It is also standard of care to continue to administer these questionnaires as symptom status changes throughout the course of treatment until discharge. At the subsequent visit, subjects will undergo cardiovascular testing on a stationary bike to identify symptom provocation and exercise tolerance with aerobic exercise. The above evaluative tools and interventions are standard of practice for concussion patients being treated by physical therapy at the Duke Sports Concussion Clinic.

Intervention Procedure (BFR):

A blood flow restriction (BFR) cuff is applied to dominant leg and limb occlusion pressure (LOP) and personalized tourniquet pressure (PTP) at 80% is determined with the patient in supine.

Using an established BFR protocol of 4 sets of exercises with repetitions of 30-15-15-15, the patient will perform the exercises of double leg squat and forward lunge under occlusion. There will be a 30 second break between each set and 1 minute break between exercises.

Then, the physical therapist will move BFR cuff to opposite leg and reassess LOP/PTP 80%. The patient will repeat squat and forward lunge exercises as above.

The treatment will be discontinued if there is a greater than 3 point change in subjective symptom report. If the patient reports leg pain/discomfort, the pressure will be decreased by 10%. If still unable to complete the exercise due to leg discomfort, the intervention will be discontinued.

The following will be recorded:

Heart rate range during each set Maximum heart rate during the recovery period Rate of Perceived Exertion (RPE) and symptom report will be obtained during each recovery period.

Total time under occlusion upon completion of the round.

Intervention Procedure (No BFR):

Subjects will perform the 4 sets of each exercise with repetitions of 30-15-15-15. There will be a 30 second break between each set and 1 minute break between exercises.

The exercises will include double leg squat, dominant leg forward lunge, repeat double leg squat, and non-dominant leg forward lunge

The following will be recorded:

Heart rate range during each set Maximum heart rate during the recovery period Rate of Perceived Exertion (RPE) and symptom report will be obtained during each recovery period.

ELIGIBILITY:
Inclusion Criteria:

Ability to read, write, and speak the English language Diagnosis of Post-Concussion Syndrome (medical diagnosis of concussion with symptoms lasting greater than four weeks.

Increased symptoms with physical activity Ages 14-30 years old

Exclusion Criteria:

Focal neurological deficits Exclusion criteria for Blood Flow Restriction (open wounds or fracture, history of clot, impaired circulation or venous compromise, sickle cell anemia, extremity infection, tumor distal to tourniquet placement, cancer, lymphectomy) Migraine history Positive image findings on MRI Benign Positional Paroxysmal Vertigo

Ages: 14 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Change in Post Concussion Symptom Score | Baseline and 8 weeks
  The Post Concussion Symptoms Score is a self-reported measurement of symptoms associated with concussion with items ranked from 0 (no symptoms) to 6 (severe symptoms)

SECONDARY OUTCOMES:
Change in Global Function Rating | Baseline and 8 weeks
  The subject will be asked to report his/her function rating on a scale of 0-100%
Change in Heart Rate Variability | 1 week, 3 weeks, 6 weeks, 8 weeks
  Heart Rate Variability will be compared, over time, to the baseline variability measured at the initial evaluation
Change in Presence of Orthostatic Tachycardia | Baseline, 1 week, 2 weeks
  Orthostatic Tachycardia will be recorded as either present or absent
Change in Presence of Orthostatic Symptoms (Headache) | Baseline, 1 week, 2 weeks
  Symptom of headache onset during a orthostatic position change will be recorded as present or not present
Change in Presence of Orthostatic Symptoms (dizziness/light headedness) | Baseline, 1 week, 2 weeks
  Symptom of dizziness/light headedness onset during a orthostatic position change will be recorded as present or absent

CONTACTS AND LOCATIONS:
Overall Officials: Laura Pietrosimone, Principal Investigator — Duke University
Locations (1):
- Duke Sports Science Institute, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No